CLINICAL TRIAL: NCT02679664
Title: StAtins for Venous Event Reduction in Patients With Venous Thromboembolism: A Pilot Study Assessing Feasibility of an RCT to Evaluate if Generic Rosuvastatin Reduces the Risk of Recurrent VTE in Patients With Symptomatic Major VTE.
Brief Title: StAtins for Venous Event Reduction in Patients With Venous Thromboembolism Pilot Study
Acronym: SAVER
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20160047-01H
Record Dates: First submitted 2016-02-01; First posted 2016-02-10 (Estimated); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment group (Experimental): 20 mg tablet of rosuvastatin PO once-a-day starting at the time of randomization until the completion of follow-up at 6 months.
  Interventions: Drug: Rosuvastatin
- Control group (No Intervention): Standard medical care only. No rosuvastatin group.

INTERVENTIONS:
Drug: Rosuvastatin — 20 mg tablet of rosuvastatin
  Other Names: Generic rosuvastatin; Teva-Rosuvastatin
  Arms: Treatment group

SUMMARY:
The SAVER pilot is a randomized, open-label pilot study to determine the feasibility of recruitment. In addition to feasibility data, the investigators will carefully collect clinical data to determine if rosuvastatin can reduce post-thrombotic syndrome (PTS) in venous thromboembolism (VTE) patients.

Eligible consenting patients who developed acute, symptomatic, and objectively confirmed proximal leg deep vein thrombosis (DVT) and/or PE will be randomized and equally allocated to 2 trial arms, either the treatment group (rosuvastatin tablet (20 mg/day) or the control group (usual care). The pilot trial consists of up to 4 study contacts over 6 months: screening, randomization, telephone follow-up (90 days), and final study visit (180 days).

DETAILED DESCRIPTION:
The SAVER pilot is a randomized, open-label pilot study to determine the feasibility of recruitment. In addition to feasibility data, the investigators will carefully collect clinical data to determine if rosuvastatin can reduce post-thrombotic syndrome (PTS) in venous thromboembolism (VTE) patients.

* SCREENING: Research coordinators at each pilot site will screen patients for eligibility and will complete detailed logs of all patients meeting inclusion (both enrolled and excluded). After providing informed consent, eligibility will be confirmed by the following tests : a lipid profile, A1C test/ CBC, transaminase (ALT) levels, Creatinine and pregnancy test (if a female of child bearing potential). Consenting participants who (following screening) do not meet eligibility criteria will be followed up to establish feasibility outcomes.
* RANDOMIZATION: Randomization will be conducted using an Interactive Web based Randomization System in a 1:1 ratio for treatment (20mg rosuvastatin od) or control (no study drug).
* STUDY DRUG DISPENSING: Participants randomized to the treatment arm will be dispensed x 200 20mg tablets of rosuvastatin along with a medication diary.They will be educated on study drug dosing regimen (20mg tablet od), how to complete their medication diary and on the possible side-effects of rosuvastatin. They will be advised to contact either the study coordinator, investigator or go directly to the emergency department should they experience any symptoms in particular anything muscle related.
* BASELINE. Assessments include;

  * Demographic data;
  * Concomitant medications (antiplatelet, anti-inflammatories, anticoagulation);
  * Type of index VTE;
  * PTS Villalta leg assessment conducted by both the participant (Patient Reported Villalta [PRV] questionnaire) and a qualified blinded independent observer (The Villalta scale is the most extensively validated tool and is recommended by the ISTH) - (Primary Outcome);
  * Risk factors for recurrent VTE, bleeding and arterial vascular events;
  * Medical history including prior VTE, Arterial disease, Liver disease and Glucose Intolerance.
* 90 DAY FOLLOW UP [Treatment arm only]: Participants randomized to treatment will be followed up via telephone or email at 90 days (+/- 21 days);

  * Participants will be asked questions to screen for;

    * Study outcomes: Suspected VTE, Arterial, Bleeding and/ or Muscle Events Patients who report any unexplained muscle symptoms will be asked to have their Creatine kinase (CK) levels tested within 2 weeks of reporting the symptoms. Study drug will be discontinued if CK levels are markedly elevated (> 10 x ULN).;
    * Study Drug compliance
    * Adverse events.
    * Concomitant medication will be reviewed in case of any contraindications. Changes or additions in concomitant anticoagulation therapy, anti-platelet or anti - inflammatory medication will also be recorded.
  * Study coordinators will log all follow up contact attempts.
* FINAL STUDY VISIT (180 days (+/- 21 days): All study participants will be asked to attend an in person study visit at 180 days (+/-21) for;

  * Follow-up of study outcomes; VTE, Arterial, Bleeding and Muscle events;
  * Study drug compliance;
  * Relevant (S)AE(s).
  * Repeat PTS leg assessment (using the Villalta scale) both by a qualified independent observer and the participant (Primary outcome);
  * Study drug compliance: Medication Diaries and used medication bottles will be collected by the study coordinator. Coordinator will perform a pill count and reconcile with the participants medication diary. Coordinator will also ask participant reasons for any missed doses.

ADJUDICATION OF STUDY OUTCOMES: All Bleeding, VTE and Arterial Suspected Events as well as deaths will be recorded on a suspected event CRF along with any diagnostic imaging/ tests and will trigger a more in-depth evaluation, and review by an independent adjudication committee.

ADVERSE EVENTS: AEs will be elicited, monitored and recorded throughout the study.

All events meeting the definition of an SAE (as per ICH-GCP) must be reported to the SAVER Trial Office in Ottawa, Canada within 24 h of awareness.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic objectively confirmed proximal leg DVT (above the trifurcation of the popliteal vein) and/or PE (segmental or greater) diagnosed in the last 30 days.

Exclusion Criteria:

1. Unable or unwilling to provide written informed consent
2. ≤ 18 years of age
3. Currently prescribed a statin
4. A medical history or current diagnosis of any of the following:

   * Abdominal aortic aneurysm,
   * Peripheral arterial disease,
   * Stroke,
   * Transient ischemic attack (TIA),
   * Myocardial infarction (MI),
   * Acute coronary syndromes,
   * Stable angina,
   * Coronary or other arterial revascularization
5. LDL-C >4.91 mmol/L
6. LDL-C between 1.81mmol/L to 4.9mmol/L AND 10 ASCVD risk score >10%
7. Diabetes mellitus or pre-diabetes
8. Contraindication to rosuvastatin;

   * Hypersensitivity or intolerance to statins;
   * History of muscle disorders or statin-related muscle pain;
   * Liver disease (active liver disease or unexplained elevations of serum transaminases exceeding 3 times the upper limit of normal);
   * Chronic kidney disease (Creatinine clearance < 30ml/min)
   * Currently pregnant or breast feeding;
   * Taking cyclosporine.
9. Life expectancy less than 3 months, as judged by the investigator
10. Unstable medical or psychological condition that would interfere with trial participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2020-01-13 (Actual); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Number of participants recruited per center per month - [Study Feasibility] | 3 years
  Study feasibility as indicated by the number of participants recruited per center per month.
Incidence of PTS | 180 days (+/- 21 days)
  Incidence of post thrombotic syndrome (PTS), as measured by the Villalta scale at 6 months by both an 'Blinded Independent Assessor' and self reported by the participant.

SECONDARY OUTCOMES:
Symptomatic recurrent major VTE | 180 days (+/- 21 days)
  Symptomatic recurrent major VTE (proximal DVT or segmental or larger PE) in patients taking generic rosuvastatin (full trial primary outcome). Coordinators will submit a report to the independent adjudication committee for participants that undergo investigation for suspected recurrent VTE during the study.
Components of major VTE | 180 days (+/- 21 days)
  1. Proximal DVT
  2. Segmental or greater PE
Non-major VTE | 180 days (+/- 21 days)
  1. Distal DVT(distal to the trifurcation of the popliteal vein)
  2. Isolated sub-segmental PE
  3. Superficial phlebitis > 5 cm
  4. Superficial phlebitis ≤ 5 cm
Arterial Vascular Events | 180 days (+/- 21 days)
  At the 3-month call and 6-month visit the research coordinator will follow an interview script to screen for inter-current suspected arterial events. Any reported potential arterial events will trigger a more in-depth evaluation.
  1. Fatal myocardial infarction
  2. Non-fatal myocardial infarction
  3. Hospitalization for unstable angina
  4. Coronary artery revascularization
  5. Sudden cardiac death
  6. Ischemic stroke
All-cause mortality | 180 days (+/- 21 days)
  All-cause mortality
Bleeding | 180 days (+/- 21 days)
  At each follow-up visit the research coordinator will follow an interview script to screen for suspected major and clinically relevant non-major bleeding events. Suspected bleeding that lasts more than 10 minutes, required intervention to control or for which the patient sought medical attention will be adjudicated by an independent committee using ISTH bleeding criteria.
Muscle Toxicity | 180 days (+/- 21 days)
  Participants reporting symptoms of muscle toxicity will have their CK levels tested for safety. Study drug will be discontinued if CK levels are markedly elevated (>10 x ULN)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Rodger, M.D., Principal Investigator — Ottawa Hospital Research Institute
Locations (6):
- Canada (5):
  - Nova Scotia Health Authority, Halifax, Nova Scotia
  - Hamilton Health Sciences Corporation, Hamilton, Ontario
  - Lawson Health Research Institute, London Health Sciences Centre, London, Ontario
  - Ottawa Hospital, Ottawa, Ontario
  - Sir Mortimer B. Davis Jewish General Hospital, Montreal, Quebec
- Østfold Hospital Trust, Grålum, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Delluc A, Ghanima W, Kovacs MJ, Shivakumar S, Kahn SR, Sandset PM, Kearon C, Mallick R, Rodger MA. Prevention of post-thrombotic syndrome with rosuvastatin: A multicenter randomized controlled pilot trial (SAVER). Thromb Res. 2022 May;213:119-124. doi: 10.1016/j.thromres.2022.03.014. Epub 2022 Mar 19. PMID 35344784